CLINICAL TRIAL: NCT01145248
Title: A Combination of Endoscopic Transpapillary Brush Cytology and a Novel Method of Forceps Biopsy to Diagnose Proximal Biliary Malignancies
Brief Title: Comparison of Biliary Forceps Biopsy and Brush Cytology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Collaborators: Heidelberg University (Other)
Responsible Party: Professor Hasan Kulaksiz, Department of Internal Medicine I, Ulm University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BilBiop_001
Record Dates: First submitted 2010-06-14; First posted 2010-06-16 (Estimated); Last update posted 2010-06-16 (Estimated); Status verified 2010-05

CONDITIONS: Cholangiocarcinoma
Keywords: Cholangiocellular Carcinoma
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Malignant biliary disease (Experimental)
  Interventions: Device: double-balloon enteroscopy forceps biopsy; Device: Transpapillary brush cytology
- Benign biliary disease (Experimental)
  Interventions: Device: double-balloon enteroscopy forceps biopsy; Device: Transpapillary brush cytology

INTERVENTIONS:
Device: double-balloon enteroscopy forceps biopsy — An endoscopic retrograde cholangiography (ERC) with a duodenoscope Olympus TFJ 160-R (Olympus Corp., Tokyo, Japan) and endoscopic sphincterotomy with an Olympus papillotome (Olympus) is performed under analgosedation . Then, the cannulation of the bile duct is performed by a pusher using a guidewire/guiding catheter. Subsequently, 2 histology samples are taken via a double-balloon enteroscopy (DBE) forceps (BF1725DF, Fujinon GmbH, Willich, Germany), which is placed under the guidance of the pusher.
Device: Transpapillary brush cytology — An endoscopic retrograde cholangiography (ERC) with a duodenoscope Olympus TFJ 160-R (Olympus Corp., Tokyo, Japan) and endoscopic sphincterotomy with an Olympus papillotome (Olympus) is performed under analgosedation . The region of interest is then brushed five times in both directions to obtain cytology specimen.

SUMMARY:
Cholangiocarcinomas (CCCs) are malignant tumors arising from the biliary epithelium. CCCs are characterised by a high mortality and the only curable therapy is complete tumor resection, if feasible, or in some cases liver transplantation. Since surgery for CCC is a procedure associated with a high mortality itself it needs to be ascertained that an accurate preoperative diagnosis has been established. However, it often appears to be difficult to get a preoperative pathological diagnosis, since it is difficult to obtain tumor specimens using cytologic brushings, biopsy forceps, bile aspiration or endoscopic ultrasonography guided-fine needle aspiration. This is reflected by a nearly 100% specificity but low sensitivity rates.

The aim of this study is to compare a new method of biliary biopsy using a double-balloon enteroscopy (DBE) forceps to enable a safe and reliable tissue specimen collection within the proximal biliary tract with cytology brushings in patients with suspected malignant proximal biliary strictures.

ELIGIBILITY:
Inclusion Criteria:

* biliary stenosis with suspected malignancy

Exclusion Criteria:

* no definite diagnosis available

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2006-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Biopsy versus brush cytology for diagnosing CCC | 6 months
  For this study we recruit patients with proximal biliary stenoses, which are suspect for malignancy. An endoscopic retrograde cholangiography (ERC) will be performed on all patients . During ERC all subjects are undergoing both biopsy (using a double-balloon enteroscopy [DBE] forceps under a guidance of a pusher and guiding catheter with guidewire) and transpapillary brush cytology. The definite clinical diagnosis will be compared to cytological/histological results obtained by biopsy/cytology and accuracy will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Kulaksiz, Professor, Principal Investigator — Department of Internal Medicine I, Ulm University Hospital
Locations (1):
- Department of Internal Medicine I, Ulm University Hospital, Ulm, Baden-Wurttemberg, Germany